CLINICAL TRIAL: NCT03719443
Title: A Phase 1, Randomized, Placebo-Controlled, Single Ascending Dose First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of VIS649 Administered Intravenously in Healthy Subjects
Brief Title: First in Human Study to Assess Safety of VIS649 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Visterra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIS649-101
Record Dates: First submitted 2018-10-10; First posted 2018-10-25 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Immunoglobulin A Nephropathy; IgAN - IgA Nephropathy; IgA Nephropathy
Keywords: chronic glomerular disease; autoimmune glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: phase 1, randomized, placebo-controlled, double-blind, single ascending dose study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The clinical study will be performed in a double-blind manner, for clinical research unit staff interacting with study participants, with the exception of the persons involved in the preparation of the IMPs. These persons will not be involved in any other study activities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VIS649 (Experimental): A single dose of VIS649 will be administered IV over approximately 1 hour on Day 1, at doses ranging from 0.5 mg/kg up to but not to exceed 20 mg/kg. No other doses will be administered during the study.
  Interventions: Biological: VIS649
- Placebo (Placebo Comparator): Single IV dose of placebo will be administered via IV over approximately 1 hour on Day 1. No other doses will be administered during the study.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VIS649 — Single IV dose of study product on Day 1 of study
  Arms: VIS649
Biological: Placebo — Singe IV dose of placebo administered via IV on Day 1 of study
  Arms: Placebo

SUMMARY:
This is a phase 1, randomized, placebo-controlled, double-blind, single ascending dose study of IV VIS649 in healthy subjects.

VIS649 is a monoclonal immunoglobulin G2 (IgG2) antibody targeting the B-cell growth factor APRILL.

The study will enroll up to 45 subjects and will be conducted in up to 5 sequential dosing cohorts at four different dose levels, enrolling 9 subjects per cohort. Subjects will be randomized to VIS649 or placebo in a ratio of 7:2 (7 active, 2 placebo). Safety, pharmacokinetic (PK) and pharmacodynamic (PD) data from the initial cohorts will be assessed.

DETAILED DESCRIPTION:
On Day 1, a single dose of VIS649 or placebo will be administered IV. Pharmacokinetics sampling will start with a collection prior to the start of infusion and at multiple timepoints throughout the study. Pharmacodynamics sampling will occur at baseline and multiple timepoints throughout the study.

Sentinel subjects will be utilized; the first two subjects in each cohort will be randomized to receive either VIS649 or placebo and will receive study drug at least 24 hours before the remaining subjects in the cohort are dosed.

The safety profile of these subjects over the 24 hour post-administration period will be reviewed to determine whether it is appropriate to proceed with enrollment of the remaining subjects in the cohort as planned. This will occur for each dose escalation.

The maximum duration of participation (Screening through End-of-study) for individual subjects will be approximately 20 weeks (5 months). The scheduled final visit will occur 16 weeks post-dosing (112 days).

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form prior to performing any of the Screening Visit procedures and be able to sign and date an appropriate Health Insurance Portability and Accountability Act (HIPAA) authorization form or subject privacy form, if appropriate.
2. Male and female subjects between 18 to 55 years of age, inclusive, at the Screening Visit.
3. For Japanese subjects: Subject is of Japanese descent as evidenced by verbal confirmation of familial heritage (a subject has all four Japanese grandparents born in Japan).
4. For non-Japanese subjects: Subjects must be of non-Asian descent, as evidenced by verbal confirmation that all four grandparents are non-Asian.
5. The following applies to female subjects:

   * Non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation]) for at least 6 months, or postmenopausal ≥ 1 year, or
   * Non-pregnant, non-lactating females of childbearing potential must report prior use (over the 28 days prior to dosing of study drug) of medically acceptable forms of birth control (hormonal contraception, abstinence, diaphragm with spermicide, condom with spermicide or intrauterine device, or partner with vasectomy), with agreement to continue to use a medically acceptable form of birth control (as described) through the end of their participation in the study. Alternatively, a reported history of abstinence beginning at least 28 days prior to study drug dosing, with agreement to continue abstinence through the end of their participation in the study are required. Females of childbearing potential must also have a negative serum human chorionic gonadotropin (hCG) pregnancy test at Screening and a negative urine hCG pregnancy test at Baseline (Day -1). Female subjects must also agree not to donate eggs/bank eggs for the duration of their participation in the study.
6. For male, subject and/or his partner must use a highly effective form of contraception (i.e., double-barrier as described above, have had a vasectomy, or have a female partner of non childbearing potential) or agree to abstinence following study drug dosing, through the end of the subject's participation in the study. Male subjects must also agree to not donate sperm for the duration of their participation in the study, following study drug dosing.
7. Screening laboratory values must meet the following criteria:

   * White blood cells 3,000 12,000/mm3
   * Platelets >150,000/mm3
   * Hemoglobin >13 gm/dL for male and>11 gm/dL for female
   * Estimated glomerular filtration rate >80 mL/min/1.73 m2
   * Serum creatinine <1.25x Upper Limit of Normal (ULN)
   * Blood Urea Nitrogen (BUN) ≤25mg/dL
   * Aspartate aminotransferase (AST) ≤50 U/L
   * Alanine aminotransferase (ALT) ≤67 U/L
   * Alkaline phosphatase ≤150 U/L
   * Total Bilirubin ≤1.4 mg/dL unless patient has Gilbert Syndrome, in which case direct bilirubin must be within normal range
   * Glucose (fasting) <115 mg/dL
   * Drug and alcohol screen Negative
   * Serum Immunoglobulin G (IgG) >750 mg/dL (7.5 g/L)
   * Serum Immunoglobulin M (IgM) >55 mg/dL (0.55 g/L)
   * Serum IgA >80 mg/dL (0.8 g/L)
8. Body mass index (BMI) between 18 and 32 kg/m2, inclusive, at the Screening Visit.
9. Healthy, determined by pre-study medical evaluation (medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations), as judged by the Investigator.
10. Is willing and able to comply with study restrictions and to remain at the central processing unit (CPU) for the in-patient duration of the study and return for all follow-up outpatient visits.
11. QTcF or QTcB < 450 msec at Screening (may be repeated once).

Exclusion Criteria:

1. Is participating in another clinical study of any investigational drug, device, or intervention or has received any investigational medication during the last 30 days or five half-lives, whichever is longer, before Baseline (Day -1).
2. Subject is judged by the Investigator or the Medical Monitor to be inappropriate for the study.
3. Subject has a history or current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, hematologic, autoimmune, blood dyscrasias or other medical disorder, including psychiatric disorders, cirrhosis or malignancy. History of minor skin cancers (not including melanoma) or surgically treated, limited cervical carcinomas (i.e., carcinoma in situ) are not exclusionary.
4. Subject has a history or presence of proteinuria, chronic kidney disease, disease requiring immunosuppressive therapy (including systemic steroids), or is considered to be immunosuppressed for any other reason.
5. Previous receipt of antibody or biologic therapy whether licensed or investigational (immunoglobulin products, monoclonal antibodies or antibody fragments) within 30 days prior to dosing or 5 half-lives within the dose of Investigational medicinal products (IMP), whichever is longer.
6. History of a previous severe allergic reaction with generalized urticaria; angioedema or anaphylaxis.
7. Blood pressure >160/100 mmHg or <90/50 mmHg (may be repeated once if abnormal), at the Screening visit and Day 1.
8. Known hypoglobulinemia disorder (i.e., common variable immunodeficiency), X linked agammaglobulinemia, selective IgA deficiency, selective IgM deficiency).
9. History of pre-existing latent infections (e.g., tuberculosis) or any infection requiring hospitalization or treatment with antivirals or antibiotics, or vaccination within 30 days prior to administration of study medication.
10. Concomitant use of marketed or investigational systemic immunosuppressive or immunomodulatory medications (e.g., corticosteroids, methotrexate, azathioprine, etc. and/or biologics) is prohibited and require a washout period prior to Screening (30 days or 5 half lives, whichever is longer).
11. Has received any prescription or non-prescription (over-the-counter [OTC]) except acetaminophen or ibuprofen, including hormonal contraceptives, topical medications, vitamins, dietary or herbal during the last 30 days or 5 half-lives, whichever is longer, preceding Baseline (Day -1).
12. Subjects who consume more than 21 units of alcohol per week (7 days) or those who have a history of alcohol or drug/chemical abuse; one unit of alcohol is equivalent to eight ounces of beer, 4 ounces of wine, or one ounce of spirits.
13. Subject is a user or former user of nicotine-containing products (including but not limited to cigarettes, cigars, and chewing or dipping tobacco) who stopped use or consumption (i.e., smoking, chewing, or pinching) of these nicotine-containing products less than 3 months before study drug administration or is using or has used topical or oral nicotine preparations for smoking cessation within the past 90 days before study drug administration.
14. Subjects who consume greater than 500 mg of caffeine or xanthine-containing products per day (e.g., coffee, tea, soft drinks, energy drinks, or chocolate).
15. Subjects who refuse to abstain from alcohol, xanthine-containing or caffeine-containing foods or beverages, or grapefruit foods or beverages, or Seville-orange containing foods (e.g., orange marmalade) or beverages, from 48 hours prior to check-in on Day-1 through the end of the study.
16. Subjects with a positive urine drug (inclusive of marijuana) or alcohol Screening test result at Screening and Day -1.
17. Subjects with a positive hepatitis B surface antigen test or evidence of chronic hepatitis C virus (HCV) infection at Screening (a negative HCV antibody assay at screening is sufficient to rule-out chronic HCV infection for this study).
18. Subjects with a known history of a positive Human Immunodeficiency Virus (HIV) or a positive test result at Screening.
19. Subjects who have donated >500 mL or blood within 60 days prior to start of Screening.
20. The subject has donated any plasma within 7 days prior to Baseline (Day -1).
21. Is an employee of the clinical research team (any Visterra or research site employee), or has a family member who is an employee of these organizations.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Yoon, MD, Principal Investigator — Parexel
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mathur M, Barratt J, Suzuki Y, Engler F, Pasetti MF, Yarbrough J, Sloan S, Oldach D. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VIS649 (Sibeprenlimab), an APRIL-Neutralizing IgG2 Monoclonal Antibody, in Healthy Volunteers. Kidney Int Rep. 2022 Feb 8;7(5):993-1003. doi: 10.1016/j.ekir.2022.01.1073. eCollection 2022 May. PMID 35570983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done for a single clinical site.
Pre-assignment Details: No notable events took place between participant enrollment and assignment.
Groups:
- Pooled Placebo: Single IV dose of placebo will be administered via IV over approximately 1 hour on Day 1.
- VIS649 Cohort 1: A single dose (0.5 mg/kg) of VIS649 administered IV over approximately 1 hour on Day 1.
- VIS649 Cohort 2: A single dose (2.0 mg/kg) of VIS649 administered IV over approximately 1 hour on Day 1.
- VIS649 Cohort 3: A single dose (6.0 mg/kg) of VIS649 administered IV over approximately 1 hour on Day 1.
- VIS649 Cohort 4: A single dose (12 mg/kg) of VIS649 administered IV over approximately 1 hour on Day 1.
- Placebo Cohort 5 + Vaccine: Single dose of placebo followed by single dose of vaccine
- VIS649 Cohort 5 + Vaccine: Single dose of 6.0 mg/kg VIS649 followed by single dose of vaccine
Period: Overall Study
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | Placebo Cohort 5 + Vaccine | VIS649 Cohort 5 + Vaccine
Started | 8 | 7 | 7 | 7 | 7 | 5 | 10
Completed | 8 | 7 | 5 | 7 | 6 | 5 | 9
Not Completed | 0 | 0 | 2 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | Placebo Cohort 5 + Vaccine | VIS649 Cohort 5 + Vaccine | Total
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 10 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (9.24) | 29.4 (6.70) | 40.4 (11.70) | 41.0 (9.63) | 40.9 (11.87) | 33.4 (8.44) | 30.9 (7.28) | 35.3 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 5 | 4 | 3 | 4 | 29
  Male | 5 | 2 | 2 | 2 | 3 | 2 | 6 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 3 | 3 | 3 | 0 | 0 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 1 | 3 | 3 | 7 | 22
  White | 1 | 2 | 1 | 3 | 1 | 2 | 3 | 13
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 7 | 7 | 7 | 5 | 10 | 51
Height (cm) [Mean (Standard Deviation); unit: cm] | 170.9 (8.22) | 165.4 (10.11) | 165.3 (11.91) | 166.4 (7.93) | 167.1 (13.04) | 167.8 (10.33) | 174.9 (11.82) | 168.7 (10.64)
Weight (kg) [Mean (Standard Deviation); unit: Kg] | 73.53 (15.378) | 69.64 (11.563) | 66.3 (16.236) | 70.03 (11.517) | 67.24 (12.699) | 71.36 (4.225) | 74.33 (10.624) | 70.60 (12.097)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.10 (4.275) | 25.39 (2.812) | 23.96 (3.625) | 24.86 (4.156) | 24.00 (2.864) | 25.52 (2.906) | 24.52 (2.011) | 24.67 (3.145)

OUTCOME MEASURES:

1. Primary Outcome: Overall Summary of Treatment Emergent Adverse Events
Description: The number adverse events (AEs), serious adverse events (SAEs), and drug related events following administration of VIS649. Safety will be assessed via AE severity per CTCAE v4.0
Time Frame: Baseline to day 112
Population: Safety Population
Measure: Number; unit: Event
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | Placebo Cohort 5 + Vaccine | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 3 | 3 | 4
Event
  Adverse Events | 8 | 3 | 7 | 7 | 7 | 6 | 4
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Drug related events | 3 | 2 | 3 | 3 | 1 | 1 | 0
  Mild severity | 4 | 2 | 2 | 1 | 3 | 3 | 4
  Moderate severity | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Severe severity | 0 | 0 | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Cmax: Maximum Serum VIS649 Concentration Determined Directly From the Concentration-time Profile. All Participants
Description: The maximum serum concentration (Cmax) of VIS649 determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. All participants
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
μg/mL | 12.600 (2.222) | 48.600 (11.660) | 135.900 (20.380) | 282.600 (48.440) | 130.700 (20.150)

3. Secondary Outcome: Tmax: Time to the Maximum Serum VIS649 Concentration Determined Directly From the Concentration-time Profile. All Participant
Description: The time to the maximum serum concentration (tmax) of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. All participants
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Median (Full Range); unit: hours
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
hours | 1.136 [1.12 to 3.11] | 3.045 [1.15 to 3.09] | 3.038 [1.13 to 3.16] | 1.148 [1.11 to 9.11] | 3.053 [1.14 to 25.11]

4. Secondary Outcome: The Pharmacokinetic Exposure Profiles of VIS649 in Serum. All Participants
Description: Summary of the pharmacokinetic profiles of VIS649 exposure in serum for all participants.
  AUC0-112 presents the area under the concentration time curve from pre-dose (time 0) to the concentration on day 112.
  AUC0-last presents the area under the concentration time curve from pre-dose (time 0) to the last quantifiable concentration.
  AUC0-inf presents the area under the concentration time curve from pre-dose (time 0) extrapolated to infinite time.
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration) including all ethnicities.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
h*μg/mL
  AUC 0-112 days | 1118 (209.4) | 11680 (3402) | 74500 (18570) | 176300 (26100) | 57900 (18390)
  AUC 0-last | 885.2 (146.2) | 10510 (2811) | 72760 (19210) | 148900 (17460) | 53630 (18180)
  AUC 0-inf | 1118 (209.5) | 11670 (3403) | 74380 (18620) | 187400 (35980) | 57910 (18390)

5. Secondary Outcome: T 1/2 The Terminal Elimination Half Life of VIS649 in Serum Samples. All Participants
Description: The terminal elimination half life (t1/2) of VIS649 from the concentration-time profile as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods.
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
hours | 60.72 (4.35) | 175.20 (38.40) | 230.90 (76.20) | 670 (179.80) | 342.10 (91.62)

6. Secondary Outcome: CL: The Clearance of VIS649 in Serum Samples Calculated Using Exposure Extrapolated to Infinity by Dose.
Description: The clearance rate (CL) of VIS649 using the exposure calculated to infinity of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. All participants.
Time Frame: Day 1 to day 112
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
mL/h | 31.46 (4.544) | 11.70 (2.522) | 6.125 (2.263) | 4.508 (1.375) | 8.724 (4.137)

7. Secondary Outcome: Vd: The Volume of Distribution of VIS649 in Serum Samples. All Participants
Description: The volume of distribution of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. All participants.
Time Frame: Day 1 to day 112
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Mean (Standard Deviation); unit: mL
Groups:
- VIS649 Cohort 5 + Vaccine: Single dose of 6.0 mg/kg VIS649 followed by single dose of TENIVAC vaccine
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
mL | 2747 (351.6) | 2854 (323.5) | 2183 (1365) | 4122 (780.4) | 3911 (828.4)

8. Secondary Outcome: Cmax: Maximum Serum VIS649 Concentration Determined Directly From the Time Profile. Japanese Participants
Description: The maximum serum concentration (Cmax) of VIS649 determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. Japanese participants
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration) of Japanese ethnicity.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
μg/mL | 11.83 (1.172) | 40.13 (4.302) | 133.0 (12.12) | 249.0 (47.84)

9. Secondary Outcome: Tmax: Time to the Maximum Serum VIS649 Concentration Determined Directly From the Concentration-time Profile. Japanese Participants
Description: The time to the maximum serum concentration (tmax) of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. Japanese participants.
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
hours | 1.136 [1.13 to 3.05] | 3.045 [1.15 to 3.09] | 3.049 [1.14 to 3.16] | 3.064 [1.12 to 9.11]

10. Secondary Outcome: The Pharmacokinetic Exposure Profiles of VIS649 in Serum. Japanese Participants
Description: AUC0-112 presents the area under the concentration time curve from pre-dose (time 0) to the concentration on day 112.
  AUC0-last presents the area under the concentration time curve from pre-dose (time 0) to the last quantifiable concentration.
  AUC0-inf presents the area under the concentration time curve from pre-dose (time 0) extrapolated to infinite time.
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration) Japanese participants.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
h*μg/mL
  AUC 0-112 days | 1039 (56.05) | 9405 (434.5) | 87210 (11210) | 185200 (32550)
  AUC 0-last | 820.6 (25.48) | 8824 (216.3) | 85750 (11220) | 150300 (21630)
  AUC 0-inf | 1039 (56.01) | 9399 (432.1) | 87170 (11210) | 203500 (47430)

11. Secondary Outcome: T1/2 The Terminal Elimination Half Life of VIS649 in Serum Samples. Japanese Participants
Description: as for outcome 5
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
hours | 59.24 (3.623) | 158.8 (14.67) | 189.8 (12.65) | 778.4 (247.3)

12. Secondary Outcome: CL: The Clearance of VIS649 in Serum Samples Calculated Using Exposure Extrapolated to Infinity by Dose. Japanese Participants
Description: The clearance rate (CL) of VIS649 using the exposure calculated to infinity of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods.
Time Frame: Day 1 to day 112.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
mL/h | 28.58 (1.794) | 12.26 (0.7651) | 4.385 (1.242) | 3.618 (1.442)

13. Secondary Outcome: Vd: The Volume of Distribution of VIS649 in Serum Samples. Japanese Participants
Description: The volume of distribution of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods.
Time Frame: Day 1 to day 112.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
mL | 2441 (197.9) | 2816 (390.3) | 1197 (344.5) | 3772 (674.7)

14. Secondary Outcome: Cmax: Maximum Serum VIS649 Concentration Determined Directly From the Concentration-time Profile. Non-Japanese Participants
Description: The maximum serum concentration (Cmax) of VIS649 determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods.
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration) of non-Japanese ethnicity.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- VIS649 Cohort 5: Single dose of 6.0 mg/kg VIS649 followed by single dose of vaccine.
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 10
μg/mL | 13.18 (2.816) | 54.95 (11.57) | 138.1 (26.80) | 307.8 (34.56) | 130.7 (20.15)

15. Secondary Outcome: Tmax: Time to the Maximum Serum VIS649 Concentration Determined Directly From the Concentration-time Profile. Non-Japanese Participants
Description: The time to the maximum serum concentration (tmax) of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods.
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 10
hours | 1.170 [1.12 to 3.11] | 2.253 [1.18 to 3.09] | 2.159 [1.13 to 3.06] | 1.142 [1.11 to 3.09] | 3.053 [1.14 to 25.11]

16. Secondary Outcome: The Pharmacokinetic Exposure Profiles of VIS649 in Serum. Non-Japanese Participants
Description: Summary of the pharmacokinetic profiles of VIS649 exposure in serum for non-Japanese participants.
  AUC0-112 presents the area under the concentration time curve from pre-dose (time 0) to the concentration on day 112.
  AUC0-last presents the area under the concentration time curve from pre-dose (time 0) to the last quantifiable concentration.
  AUC0-inf presents the area under the concentration time curve from pre-dose (time 0) extrapolated to infinite time.
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration) non-Japanese participants.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 10
h*μg/mL
  AUC 0-112 days | 1177 (273.4) | 13380 (3741) | 64960 (17990) | 169700 (22790) | 57900 (18390)
  AUC 0-last | 933.6 (187.1) | 11780 (3283) | 63020 (18950) | 147900 (17160) | 53630 (18180)
  AUC 0-inf | 1177 (273.6) | 13380 (3741) | 64790 (17980) | 175300 (25200) | 57910 (18390)

17. Secondary Outcome: T1/2 The Terminal Elimination Half Life of VIS649 in Serum Samples. Non-Japanese Participants
Description: The terminal elimination half life (t1/2) of VIS649 from the concentration-time profile as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. Non-Japanese participants.
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 10
hours | 61.83 (5.017) | 187.6 (48.26) | 261.8 (92.45) | 588.8 (57.65) | 342.1 (91.62)

18. Secondary Outcome: CL: The Clearance of VIS649 in Serum Samples Calculated Using Exposure Extrapolated to Infinity by Dose. Non-Japanese Participants
Description: as for outcome 12
Time Frame: Day 1 to day 112.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 10
mL/h | 33.63 (4.959) | 11.27 (3.431) | 7.430 (1.978) | 5.175 (1.004) | 8.724 (4.137)

19. Secondary Outcome: Vd: The Volume of Distribution of VIS649 in Serum Samples. Non-Japanese Participants
Description: as for outcome 13
Time Frame: Day 1 to day 112.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 10
mL | 2976 (241.0) | 2882 (324.3) | 2923 (1395) | 4384 (837) | 3911 (828.4)

20. Secondary Outcome: Pharmacodynamic Effect of VIS649 on Total Immunoglobulin G Species. All Participants
Description: The effect of VIS649 treatment on total IgG levels in serum, weekly observations from baseline to Week 24
Time Frame: From baseline to Week 24
Population: Pharmacodynamic population: the Safety Population subset with at least 1 pharmacodynamic parameter assessment post study drug dosing.
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | Placebo Cohort 5 + Vaccine | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 10
mg/dL
  Baseline | 1138.0 (288.08) | 1057 (276.8) | 1243 (293.55) | 1239.0 (269.73) | 1125.0 (262.83) | 1080.0 (225.92) | 1143.0 (213.59)
  Week 1 | 1152.0 (323.58) | 1028.0 (257.12) | 1140.0 (212.10) | 1142.0 (246.84) | 1174.0 (298.25) | 1098.0 (225.06) | 1092.5 (263.15)
  Week 2 | 1150.5 (280.89) | 987.0 (271.89) | 1120.0 (220.63) | 1108.0 (196.16) | 1038.0 (240.46) | 1117.0 (201.08) | 1053.5 (216.66)
  Week 3 | 1174.0 (293.55) | 946.0 (242.33) | 1077.0 (214.35) | 1076 (214.49) | 999.0 (212.58) | 1063.0 (202.43) | 966.5 (235.63)
  Week 4: number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 9
  Week 4 | 1184.0 (304.93) | 1122.0 (264.19) | 1038.0 (218.35) | 1053.0 (196.39) | 1034 (221.08) | 1077.0 (186.74) | 1050.0 (204.29)
  Week 5: number analyzed (Participants) | 8 | 7 | 6 | 7 | 7 | 5 | 9
  Week 5 | 1143.5 (237.34) | 994.0 (276.89) | 965.0 (193.19) | 1005.0 (216.24) | 980.0 (184.59) | 1094.0 (180.03) | 962.0 (197.14)
  Week 6: number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 9
  Week 6 | 1185.5 (295.65) | 1105.0 (285.27) | 990.0 (216.58) | 1001.0 (212.64) | 850.0 (191.40) | 1111.0 (202.60) | 971.0 (194.19)
  Week 7: number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 0 | 0
  Week 7 | 1195.0 (296.0) | 950.5 (320.91) | 1005.0 (236.55) | 948.0 (195.02) | 929.0 (184.67) |  |
  Week 8: number analyzed (Participants) | 8 | 6 | 6 | 7 | 6 | 5 | 9
  Week 8 | 1199.5 (311.20) | 1022.0 (287.47) | 1022.5 (220.65) | 974.0 (174.83) | 951.5 (222.49) | 1117.0 (223.8) | 953.0 (192.19)
  Week 10: number analyzed (Participants) | 8 | 7 | 5 | 7 | 7 | 5 | 9
  Week 10 | 1266.0 (301.04) | 1035.0 (333.11) | 985.0 (234.14) | 1006.0 (223.84) | 841.0 (196.81) | 1037.0 (196.39) | 845.0 (211.71)
  Week 12: number analyzed (Participants) | 8 | 7 | 5 | 6 | 7 | 5 | 9
  Week 12 | 1215.0 (282.42) | 992.0 (287.94) | 1036.0 (238.29) | 1027.0 (168.63) | 718.0 (185.80) | 1101.0 (205.66) | 970.0 (256.28)
  Week 14: number analyzed (Participants) | 8 | 7 | 5 | 6 | 7 | 0 | 0
  Week 14 | 1180.0 (282.87) | 1038.0 (278.83) | 930.0 (268.00) | 1071.5 (160.55) | 862.0 (180.07) |  |
  Week 16: number analyzed (Participants) | 8 | 7 | 5 | 7 | 7 | 5 | 9
  Week 16 | 1147.5 (278.04) | 1072.0 (242.20) | 934.0 (356.27) | 1104.0 (233.23) | 876.0 (220.38) | 1198.0 (156.10) | 1049.0 (261.94)
  Week 20: number analyzed (Participants) | 8 | 0 | 0 | 7 | 7 | 0 | 0
  Week 20 | 1269.0 (279.38) |  |  | 1089.0 (260.55) | 1009.0 (243.52) |  |
  Week 24: number analyzed (Participants) | 8 | 0 | 0 | 7 | 7 | 0 | 0
  Week 24 | 1250.5 (312.89) |  |  | 1075.0 (260.55) | 917.5 (91.00) |  |

21. Secondary Outcome: Pharmacodynamic Effect of VIS649 on Total Immunoglobulin A Species. All Participants
Description: The effect of VIS649 treatment on total IgA levels in serum, weekly observations from Baseline to Week 24
Time Frame: From baseline to Week 24
Population: as for outcome 20
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | Placebo Cohort 5 + Vaccine | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 10
mg/dL
  Baseline | 217.0 (70.44) | 202.0 (71.69) | 213.0 (82.89) | 233.0 (136.30) | 243.0 (96.48) | 202.0 (77.00) | 222.5 (65.16)
  Week 1 | 225.0 (68.74) | 165.0 (64.10) | 223.0 (64.03) | 209.0 (120.23) | 214.0 (100.42) | 198.0 (84.45) | 205.5 (57.03)
  Week 2 | 222.5 (74.97) | 151.0 (60.23) | 168.0 (52.76) | 187.0 (111.5) | 174.0 (82.09) | 205.0 (83.70) | 179.0 (48.79)
  Week 3 | 217.0 (73.17) | 147.0 (54.07) | 158.0 (49.15) | 163.0 (103.95) | 155.0 (74.91) | 193.0 (84.93) | 155.5 (41.48)
  Week 4: number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 9
  Week 4 | 227.0 (76.14) | 169.0 (75.99) | 134.0 (48.87) | 152.0 (87.08) | 146.0 (73.05) | 197.0 (81.96) | 150.0 (42.75)
  Week 5: number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 9
  Week 5 | 208.5 (71.81) | 164.0 (64.44) | 133.0 (43.46) | 142.0 (87.7) | 128.0 (60.93) | 194.0 (87.73) | 137.0 (38.30)
  Week 6: number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 9
  Week 6 | 217.5 (71.98) | 167.0 (67.82) | 140.0 (51.43) | 134.0 (76.69) | 116.0 (66.61) | 207.0 (90.44) | 129.0 (37.00)
  Week 7: number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 0 | 0
  Week 7 | 229.0 (68.86) | 152.5 (71.68) | 148.0 (53.76) | 113.0 (74.53) | 110.5 (68.99) |  |
  Week 8: number analyzed (Participants) | 8 | 6 | 6 | 7 | 6 | 5 | 9
  Week 8 | 217.0 (68.26) | 159.5 (74.21) | 148.5 (59.02) | 109.0 (68.40) | 111.0 (66.42) | 210.0 (92.31) | 122.0 (35.26)
  Week 10: number analyzed (Participants) | 8 | 7 | 5 | 7 | 7 | 5 | 9
  Week 10 | 215.5 (67.79) | 161.0 (59.74) | 171.0 (60.80) | 123.0 (89.55) | 105.0 (61.87) | 207.0 (83.97) | 127.0 (46.87)
  Week 12: number analyzed (Participants) | 8 | 7 | 5 | 6 | 7 | 5 | 9
  Week 12 | 227.5 (74.44) | 169.0 (65.26) | 171.0 (59.46) | 179.0 (107.20) | 87.0 (59.27) | 192.0 (85.87) | 144.0 (54.34)
  Week 14: number analyzed (Participants) | 8 | 7 | 5 | 6 | 7 | 0 | 0
  Week 14 | 232.0 (69.85) | 182.0 (70.26) | 164.0 (63.82) | 195.5 (105.85) | 109.0 (56.66) |  |
  Week 16: number analyzed (Participants) | 8 | 7 | 5 | 7 | 7 | 5 | 9
  Week 16 | 220.0 (70.88) | 179.0 (69.35) | 165.0 (89.38) | 158.0 (116.54) | 124.0 (71.96) | 192.0 (85.98) | 169.0 (52.57)
  Week 20: number analyzed (Participants) | 4 | 0 | 0 | 7 | 7 | 0 | 0
  Week 20 | 243.5 (90.16) |  |  | 172.0 (117.30) | 153.0 (67.43) |  |
  Week 24: number analyzed (Participants) | 4 | 0 | 0 | 7 | 6 | 0 | 0
  Week 24 | 239.0 (94.36) |  |  | 164.0 (123.92) | 153.5 (83.43) |  |

22. Secondary Outcome: Pharmacodynamic Effect of VIS649 on Total Immunoglobulin M Species. All Participants
Description: The effect of VIS649 treatment on total IgM levels in serum, weekly observations from Baseline to Week 24
Time Frame: From baseline to Week 24
Population: as for outcome 20
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | Placebo Cohort 5 + Vaccine | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 10
mg/dL
  Baseline | 105.0 (43.75) | 116.0 (42.77) | 93.0 (61.79) | 108.0 (49.11) | 133.0 (31.67) | 85.0 (35.75) | 132.0 (34.80)
  Week 1 | 108.0 (38.78) | 117.0 (39.91) | 70.0 (46.31) | 100.0 (46.15) | 128.0 (28.80) | 85.0 (36.02) | 102.5 (31.82)
  Week 2 | 109.5 (42.39) | 91.0 (39.04) | 58.0 (38.17) | 88.0 (43.68) | 94.0 (29.89) | 87.0 (30.86) | 87.0 (25.15)
  Week 3 | 105.0 (39.49) | 85.0 (34.49) | 52.0 (35.40) | 71.0 (38.17) | 80.0 (26.13) | 86.0 (38.91) | 73.5 (24.02)
  Week 4: number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 9
  Week 4 | 107.5 (43.13) | 84.0 (40.45) | 46.0 (31.08) | 58.0 (34.95) | 75.0 (25.32) | 81.0 (35.91) | 68.0 (20.35)
  Week 5: number analyzed (Participants) | 8 | 7 | 6 | 7 | 7 | 5 | 9
  Week 5 | 106.0 (39.41) | 83.0 (34.54) | 40.5 (23.01) | 49.0 (32.13) | 60.0 (19.85) | 84.0 (35.50) | 54.0 (15.41)
  Week 6: number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 9
  Week 6 | 106.5 (42.10) | 92.0 (37.21) | 46.0 (30.33) | 49 (30.35) | 57.0 (21.07) | 90 (35.22) | 48.0 (13.30)
  Week 7: number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 0 | 0
  Week 7 | 109.5 (44.41) | 86.5 (35.07) | 48.0 (31.14) | 43.0 (23.88) | 51.5 (18.5) |  |
  Week 8: number analyzed (Participants) | 8 | 6 | 6 | 7 | 6 | 5 | 9
  Week 8 | 110.5 (40.73) | 89.5 (37.91) | 43.0 (26.77) | 46.0 (23.80) | 46.0 (19.31) | 89.0 (33.93) | 42.0 (11.07)
  Week 10: number analyzed (Participants) | 8 | 7 | 5 | 7 | 7 | 5 | 9
  Week 10 | 104.5 (40.87) | 106.0 (40.44) | 53.0 (29.95) | 49.0 (25.15) | 44.0 (18.09) | 80.0 (32.38) | 49.0 (19.53)
  Week 12: number analyzed (Participants) | 8 | 7 | 5 | 6 | 7 | 5 | 9
  Week 12 | 113.0 (41.39) | 106.0 (37.89) | 54.0 (36.41) | 73.5 (26.46) | 35.0 (20.30) | 93.0 (41.37) | 63.0 (25.09)
  Week 14: number analyzed (Participants) | 8 | 7 | 5 | 6 | 7 | 0 | 0
  Week 14 | 113.0 (40.09) | 114.0 (41.32) | 55.0 (33.05) | 82.5 (30.31) | 44.0 (15.14) |  |
  Week 16: number analyzed (Participants) | 8 | 7 | 5 | 7 | 7 | 5 | 9
  Week 16 | 107.0 (40.51) | 127.0 (40.51) | 60.0 (30.70) | 78.0 (39.52) | 55.0 (24.08) | 93.0 (31.11) | 87.0 (30.55)
  Week 20: number analyzed (Participants) | 4 | 0 | 0 | 7 | 7 | 0 | 0
  Week 20 | 80.0 (42.54) |  |  | 90.0 (38.11) | 69.0 (23.84) |  |
  Week 24: number analyzed (Participants) | 4 | 0 | 0 | 7 | 6 | 0 | 0
  Week 24 | 89.0 (33.56) |  |  | 89.0 (40.15) | 74.5 (21.08) |  |

23. Secondary Outcome: Pharmacodynamic Effect of VIS649 on Circulating CD16 +CD56 (Natural Killer) Cells for All Participants in Cohorts 1-4
Description: The effect of VIS649 treatment on the population of circulating CD16 +CD56 (Natural killer) cells in serum for all participants in cohorts 1-4.
Time Frame: From baseline to Week 24
Population: as for outcome 20
Measure: Median (Standard Deviation); unit: cells/mcl
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7
cells/mcl
  Baseline | 122.0 (156.14) | 136.0 (38.34) | 174.0 (88.43) | 107.0 (40.82) | 142.0 (48.32)
  Week 4: number analyzed (Participants) | 8 | 5 | 7 | 7 | 7
  Week 4 | 142.5 (136.42) | 103.0 (46.6) | 144.0 (46.13) | 143.0 (45.80) | 181.0 (82.05)
  Week 16: number analyzed (Participants) | 7 | 7 | 5 | 7 | 7
  Week 16 | 130.0 (30.41) | 150.0 (34.55) | 226.0 (90.19) | 138.0 (49.69) | 153.0 (54.99)
  Week 20: number analyzed (Participants) | 4 | 0 | 0 | 7 | 7
  Week 20 | 204.0 (201.87) |  |  | 181.0 (58.45) | 189.0 (120.94)
  Week 24: number analyzed (Participants) | 4 | 0 | 0 | 7 | 5
  Week 24 | 195.0 (173.776) |  |  | 135.0 (41.35) | 270.0 (142.83)

24. Secondary Outcome: Pharmacodynamic Effect of VIS649 on Circulating CD19 (B Cells) for All Participants in Cohorts 1-4
Description: The effect of VIS649 treatment on the population of circulating CD19 (B Cells) in serum for all participants in cohorts 1-4.
Time Frame: From baseline to Week 24
Population: as for outcome 20
Measure: Median (Standard Deviation); unit: cells/uL
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7
cells/uL
  Baseline | 165 (128.25) | 193.0 (23.72) | 244.0 (89.67) | 268.0 (79.96) | 179.0 (49.44)
  Week 4: number analyzed (Participants) | 8 | 5 | 7 | 7 | 7
  Week 4 | 187.0 (73.92) | 206.0 (34.69) | 204.0 (78.55) | 294.0 (129.97) | 202.0 (67.12)
  Week 16: number analyzed (Participants) | 7 | 7 | 5 | 7 | 7
  Week 16 | 166.0 (93.65) | 226.0 (51.84) | 209.0 (98.99) | 359.0 (113.22) | 167.0 (55.86)
  Week 20: number analyzed (Participants) | 4 | 0 | 0 | 7 | 7
  Week 20 | 277.5 (70.72) |  |  | 320.0 (146.34) | 190.0 (72.04)
  Week 24: number analyzed (Participants) | 4 | 0 | 0 | 7 | 5
  Week 24 | 270.5 (76.49) |  |  | 267.0 (65.38) | 239.0 (76.41)

25. Secondary Outcome: Pharmacodynamic Effect of VIS649 on Circulating CD4 T Cells for All Participants in Cohorts 1-4
Description: The effect of VIS649 treatment on the population of circulating CD4 T cells in serum for all participants in cohorts 1-4.
Time Frame: From baseline to Week 24
Population: as for outcome 20
Measure: Median (Standard Deviation); unit: cells/uL
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7
cells/uL
  Baseline | 679.0 (178.00) | 592.0 (156.93) | 755.0 (145.8) | 553.0 (288.67) | 698.0 (166.09)
  Week 4: number analyzed (Participants) | 8 | 5 | 7 | 7 | 7
  Week 4 | 601.5 (91.92) | 631.0 (182.52) | 733.0 (194.08) | 592.0 (337.55) | 813.0 (233.06)
  Week 16: number analyzed (Participants) | 7 | 7 | 5 | 7 | 7
  Week 16 | 608.0 (153.29) | 649.0 (198.87) | 718 (127.74) | 606.0 (347.79) | 799.0 (208.09)
  Week 20: number analyzed (Participants) | 4 | 0 | 0 | 7 | 7
  Week 20 | 895.0 (279.84) |  |  | 630.0 (300.58) | 738.0 (255.19)
  Week 24: number analyzed (Participants) | 4 | 0 | 0 | 7 | 5
  Week 24 | 917.0 (245.42) |  |  | 499.0 (196.44) | 992.0 (374.77)

26. Secondary Outcome: Pharmacodynamic Effect of VIS649 on Circulating CD3 T Cells for All Participants in Cohorts 1-4
Description: The effect of VIS649 treatment on the population of circulating CD3 T cells in serum for all participants in cohorts 1-4.
Time Frame: From baseline to Week 24
Population: as for outcome 20
Measure: Median (Standard Deviation); unit: cells/uL
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7
cells/uL
  Baseline | 1147.5 (313.07) | 1118.0 (284.46) | 1218.0 (200.20) | 985.0 (365.33) | 991.0 (318.12)
  Week 4: number analyzed (Participants) | 8 | 5 | 7 | 7 | 7
  Week 4 | 1074.0 (186.09) | 993.0 (292.84) | 1110.0 (358.19) | 1018.0 (407.5) | 1226.0 (433.57)
  Week 16: number analyzed (Participants) | 7 | 7 | 5 | 7 | 7
  Week 16 | 1025.0 (300.38) | 1085.0 (220.178) | 1082.0 (140.94) | 1208.0 (437.35) | 1270.0 (367.31)
  Week 20: number analyzed (Participants) | 4 | 0 | 0 | 7 | 7
  Week 20 | 1565.0 (340.67) |  |  | 970.0 (387.46) | 1139.0 (558.77)
  Week 24: number analyzed (Participants) | 4 | 0 | 0 | 7 | 5
  Week 24 | 1644.5 (299.56) |  |  | 868.0 (207.34) | 1259.0 (722.50)

27. Secondary Outcome: Pharmacodynamic Effect of VIS649 on Circulating CD8 T Cells for All Participants in Cohorts 1-4
Description: The effect of VIS649 treatment on the population of circulating CD8 T cells in serum for all participants in cohorts 1-4.
Time Frame: From baseline to Week 24
Population: as for outcome 20
Measure: Median (Standard Deviation); unit: cells/uL
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7
cells/uL
  Baseline | 483.5 (145.06) | 442.0 (165.29) | 356.0 (103.21) | 373.0 (108.08) | 327 (199.67)
  Week 4: number analyzed (Participants) | 8 | 5 | 7 | 7 | 7
  Week 4 | 424.0 (112.24) | 338.0 (135.81) | 373.0 (152.41) | 370.0 (129.55) | 397.0 (246.05)
  Week 16: number analyzed (Participants) | 7 | 7 | 5 | 7 | 7
  Week 16 | 373.0 (166.71) | 471.0 (66.20) | 349.0 (66.96) | 391.0 (137.52) | 461.0 (210.56)
  Week 20: number analyzed (Participants) | 4 | 0 | 0 | 7 | 7
  Week 20 | 623.0 (110.15) |  |  | 362.0 (145.02) | 416.0 (359.67)
  Week 24: number analyzed (Participants) | 4 | 0 | 0 | 7 | 5
  Week 24 | 702.0 (86.56) |  |  | 322.0 (66.27) | 342.0 (443.94)

28. Secondary Outcome: Summary of Anti -VIS649 Anti-drug Antibodies (ADA)
Description: Summary of Anti -VIS649 anti-drug antibodies (ADA) by treatment group, all participants
Time Frame: Baseline to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | Placebo Cohort 5 + Vaccine | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 10
Participants
  Baseline: Negative | 8 | 7 | 7 | 7 | 7 | 5 | 10
  Baseline: Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 8 | 7 | 7 | 7 | 7 | 5 | 9
  Week 4: Negative | 8 | 7 | 7 | 7 | 7 | 5 | 8
  Week 4: Positive | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Week 8: number analyzed (Participants) | 8 | 6 | 6 | 7 | 6 | 5 | 9
  Week 8: Negative | 8 | 6 | 5 | 7 | 6 | 5 | 8
  Week 8: Positive | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Week 16: number analyzed (Participants) | 8 | 7 | 5 | 7 | 7 | 5 | 9
  Week 16: Negative | 8 | 7 | 3 | 5 | 3 | 5 | 7
  Week 16: Positive | 0 | 0 | 2 | 2 | 4 | 0 | 2

29. Secondary Outcome: Summary of Anti -VIS649 Antibody (ADA) Titer by Treatment
Description: Summary of Anti -VIS649 antibody (ADA) titer by treatment, all participants with ADA positive results
Time Frame: Baseline to Day 112
Population: Safety Population
Measure: Median (Standard Deviation); unit: titer
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | Placebo Cohort 5 + Vaccine | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 0 | 0 | 3 | 2 | 4 | 0 | 4
titer
  Week 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Week 4 |  |  |  |  |  |  | 1.0
  Week 8: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Week 8 |  |  | 0.0 |  |  |  | 0.0
  Week 16: number analyzed (Participants) | 0 | 0 | 2 | 2 | 4 | 0 | 2
  Week 16 |  |  | 32.0 (45.25) | 18.0 (19.80) | 6.0 (6.83) |  | 2.0 (2.83)

30. Secondary Outcome: Cmax: Maximum Serum VIS649 Concentration Determined Directly From the Concentration-time Profile. All Participants by Anti-VIS649 Status
Description: The maximum serum concentration (Cmax) of VIS649 determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. All participants by anti-VIS649 status (positive or negative).
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
μg/mL
  Negative: number analyzed (Participants) | 7 | 5 | 5 | 3 | 7
  Negative | 12.600 (2.222) | 48.660 (12.040) | 134.100 (23.730) | 259.000 (65.110) | 136.300 (18.420)
  Positive: number analyzed (Participants) | 0 | 2 | 2 | 4 | 3
  Positive |  | 48.450 (15.340) | 140.500 (13.440) | 300.300 (29.900) | 117.700 (21.140)

31. Secondary Outcome: Tmax: Time to the Maximum Serum VIS649 Concentration Determined Directly From the Concentration-time Profile. All Participants by Anti-VIS649 Status
Description: The time to the maximum serum concentration (tmax) of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. All participants by anti-VIS649 status (positive or negative).
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Median (Full Range); unit: hours
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
hours
  Negative: number analyzed (Participants) | 7 | 5 | 5 | 3 | 7
  Negative | 1.136 [1.12 to 3.11] | 1.434 [1.15 to 3.09] | 3.038 [1.14 to 3.16] | 3.064 [1.11 to 9.11] | 3.049 [1.14 to 25.11]
  Positive: number analyzed (Participants) | 0 | 2 | 2 | 4 | 3
  Positive |  | 3.058 [3.05 to 3.07] | 2.089 [1.13 to 3.05] | 1.142 [1.12 to 3.09] | 3.055 [3.05 to 3.07]

32. Secondary Outcome: The Pharmacokinetic Exposure Profiles of VIS649 in Serum Samples, All Participants by Anti-VIS649 Antibody Status.
Description: Summary of the pharmacokinetic profiles of VIS649 exposure in serum for all participants based on their anti-VIS649 antibody status (negative/positive).
  AUC0-112 presents the area under the concentration time curve from pre-dose (time 0) to the concentration on day 112.
  AUC0-last presents the area under the concentration time curve from pre-dose (time 0) to the last quantifiable concentration.
  AUC0-inf presents the area under the concentration time curve from pre-dose (time 0) extrapolated to infinite time.
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
h*μg/mL
  AUC 0-112 days--ADA Negative participants: number analyzed (Participants) | 7 | 5 | 5 | 3 | 7
  AUC 0-112 days--ADA Negative participants | 1118 (209.400) | 12270 (3876) | 71440 (19090) | 177700 (31330) | 56390 (17870)
  AUC 0-112 days--ADA Positive participants: number analyzed (Participants) | 0 | 2 | 2 | 4 | 3
  AUC 0-112 days--ADA Positive participants |  | 10200 (1805) | 82120 (21210) | 175300 (26540) | 61450 (23170)
  AUC 0-last--ADA negative participants: number analyzed (Participants) | 7 | 5 | 5 | 3 | 7
  AUC 0-last--ADA negative participants | 885.2 (146.200) | 10750 (3277) | 69700 (20050) | 145100 (16950) | 51550 (17860)
  AUC 0-last--ADA positive participants: number analyzed (Participants) | 0 | 2 | 2 | 4 | 3
  AUC 0-last--ADA positive participants |  | 9922 (1863) | 80410 (21040) | 151800 (19810) | 58500 (21880)
  AUC 0-inf--ADA negative participants: number analyzed (Participants) | 7 | 5 | 5 | 3 | 7
  AUC 0-inf--ADA negative participants | 1118 (209.500) | 12260 (3878) | 71340 (19120) | 194300 (49280) | 56450 (17930)
  AUC 0-inf--ADA positive participants: number analyzed (Participants) | 0 | 2 | 2 | 4 | 3
  AUC 0-inf--ADA positive participants |  | 10200 (1806) | 81980 (21350) | 182100 (29760) | 61320 (23060)

33. Secondary Outcome: T1/2 The Terminal Elimination Half Life of VIS649 in Serum Samples. All Participants by Anti-VIS649 Antibody Status.
Description: The terminal elimination half life (t1/2) of VIS649 from the concentration-time profile as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. All participants by anti-VIS649 antibody status (negative/positive).
Time Frame: 0, 1, 2, 8, and 24-hours post-dose, Day 3, 7, 14, 28, 42, 56, 70, and 112.
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
hours
  T1/2 ADA Negative participants: number analyzed (Participants) | 7 | 5 | 5 | 3 | 7
  T1/2 ADA Negative participants | 60.720 (4.346) | 192.600 (29.040) | 224.600 (85.810) | 738.4 (281.800) | 335.300 (96.780)
  T1/2 ADA Positive participants: number analyzed (Participants) | 0 | 2 | 2 | 4 | 3
  T1/2 ADA Positive participants |  | 131.900 (14.750) | 246.600 (68.520) | 618.8 (59.450) | 358.200 (95.520)

34. Secondary Outcome: CL: The Clearance of VIS649 in Serum Samples Calculated Using Exposure Extrapolated to Infinity by Dose. All Participants by Anti-VIS649 Antibody Status.
Description: The clearance rate (CL) of VIS649 using the exposure calculated to infinity of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. All participants by anti-VIS649 antibody status (positive or negative)..
Time Frame: 112 days
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
mL/h
  CL--ADA negative participants: number analyzed (Participants) | 7 | 5 | 5 | 3 | 7
  CL--ADA negative participants | 31.460 (4.544) | 10.870 (2.023) | 6.536 (2.203) | 4.019 (1.500) | 9.272 (4.765)
  CL--ADA positive participants: number analyzed (Participants) | 0 | 2 | 2 | 4 | 3
  CL--ADA positive participants |  | 13.750 (3.153) | 5.097 (2.890) | 4.875 (1.364) | 7.445 (2.324)

35. Secondary Outcome: Vd: The Volume of Distribution of VIS649 in Serum Samples. All Participants by Anti-VIS649 Antibody Status (Positive or Negative)
Description: The calculated volume of distribution of VIS649 as determined by an electrochemiluminescence (ECL) immunoassay and analyzed by standard non-compartmental pharmacokinetic methods. All participants by anti-VIS649 antibody status (positive or negative).
Time Frame: 112 days
Population: Pharmacokinetic Population (all randomized participants with at least 1 quantifiable VIS649 concentration).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | VIS649 Cohort 5 + Vaccine
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 10
mL
  Vd--ADA negative: number analyzed (Participants) | 7 | 5 | 5 | 3 | 7
  Vd--ADA negative | 2747 (351.600) | 2961 (287.200) | 2274 (1474) | 3894 (548.8) | 4026 (983.8)
  Vd--ADA positive: number analyzed (Participants) | 0 | 2 | 2 | 4 | 3
  Vd--ADA positive |  | 2584 (307.500) | 1956 (1532) | 4292 (962.6) | 3641 (171.100)

ADVERSE EVENTS:
Time Frame: From Day -1 to Day 112
Description: Standard definitions of adverse and serious adverse event were used. Severity was either mild, moderate or severe as determined by the investigator using standard criteria in the protocol. All participants were monitored in the clinic for 24 hours post dose. Additional clinical visits occurred on days 3, 7, 14, 21, 28, 35, 42, 49, 56, 70, 84, 98, 112.
Arm/Group | Pooled Placebo | VIS649 Cohort 1 | VIS649 Cohort 2 | VIS649 Cohort 3 | VIS649 Cohort 4 | Placebo Cohort 5 + Vaccine | VIS649 Cohort 5 + Vaccine
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/7 | 0/7 | 0/7 | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7 | 0/7 | 0/7 | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 4/8 | 2/7 | 3/7 | 3/7 | 3/7 | 3/5 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=8) | VIS649 Cohort 1 (N=7) | VIS649 Cohort 2 (N=7) | VIS649 Cohort 3 (N=7) | VIS649 Cohort 4 (N=7) | Placebo Cohort 5 + Vaccine (N=5) | VIS649 Cohort 5 + Vaccine (N=10)
Diarrhoea, Food poisoning, Constipation, or Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
General disorders and administration site conditions (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dizziness, Headache, Head discomfort, Migraine, Somnolence, Syncope, or Taste disorder (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain or Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain or Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Protocol Amendment 2 (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03719443/Prot_000.pdf
  • Study Protocol: Protocol Amendment 1 (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT03719443/Prot_001.pdf
  • Study Protocol: Final Protocol (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT03719443/Prot_002.pdf
  • Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT03719443/SAP_003.pdf